CLINICAL TRIAL: NCT00353301
Title: A Phase II Single Arm Clinical Trial to Evaluate the Efficacy and Safety of the Combination of Tarceva™ (Erlotinib Hydrochloride) and Rapamune™ (Sirolimus) in the Treatment of Metastatic Renal Cell Carcinoma.
Brief Title: Erlotinib and Sirolimus for the Treatment of Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-1135.cc
Record Dates: First submitted 2006-07-14; First posted 2006-07-18 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Renal Cell Carcinoma
Keywords: Carcinoma, Renal Cell; Receptor, Epidermal Growth Factor; mTOR protein; Sirolimus; Erlotinib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Erlotinib Hydrochloride; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib and Sirolimus (Experimental): Erlotinib hydrochloride (Tarceva) will be self-administered in an open-label unblinded manner to all patients enrolled in the study. During the treatment period, patients will receive single-agent Tarceva, 150 mg/day.
  Sirolimus (Rapamune) will be self-administered in an open-label unblinded manner to all patients enrolled in the study. Patients will receive a loading dose of 6 mg of Rapamune seven days after beginning treatment with Tarceva™ followed by a dose of 2mg/day.
  Interventions: Drug: Erlotinib hydrochloride; Drug: Sirolimus

INTERVENTIONS:
Drug: Erlotinib hydrochloride — Patients will receive single-agent Tarceva, 150 mg/day
  Other Names: Tarceva
Drug: Sirolimus — Patients will receive a loading dose of 6 mg of Rapamune seven days after beginning treatment with Tarceva™ followed by a dose of 2mg/day.
  Other Names: Rapamune

SUMMARY:
The purpose of this study is to test the safety and efficacy of the combination of erlotinib hydrochloride (Tarceva™) and sirolimus (Rapamune™) in the treatment of patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
Despite recent advances metastatic renal cell carcinoma remains an incurable condition. Currently available treatment with high-dose interleukin-2 can lead to complete responses in a small minority of selected patients but is markedly toxic and not broadly available. FDA-approved multikinase inhibitors (sorafenib and sunitinib malate) often cause partial and transient tumor regression. There is no standard treatment metastatic renal cell carcinoma for patients whose disease progressed on multikinase inhibitors. The kinase mammalian target of rapamycin (mTOR) is overstimulated in a subset of renal cell carcinomas and other malignancies and can be blocked by sirolimus leading to growth arrest. Erlotinib hydrochloride is a drug that blocks the function of the epidermal growth factor receptor (EGFR), often over expressed in kidney cancer. Sirolimus and EGFR inhibitors and been safely used in combination. In vitro experiments show that erlotinib enhances the sirolimus induced growth impairment in a panel of renal cell carcinoma cells. In the present study patients with metastatic renal cell carcinoma whose disease progressed on multikinase inhibitors will be treated with the combination of erlotinib hydrochloride (Tarceva™) and sirolimus (Rapamune™). This is a single arm trial with no placebo or drug-based control arm

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in this study.
* Histological diagnosis of renal cell carcinoma.
* Age greater or equal 18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance status of 2 or better.
* Life expectancy of at least 3 months.
* Failure or intolerance to previous treatment with Sutent® and/or Nexavar®.
* Most recent systemic treatment at least 1 month from the beginning of treatment.
* Most recent local treatment (surgery or irradiation) > 2 weeks from the beginning of treatment.
* At least one site of measurable disease by CT scan or MRI (RECIST criteria).
* Baseline hemoglobin >9 g/dl, platelets > 100,000/mm3, absolute neutrophil count (ANC >1500/mm3.

Exclusion Criteria:

* Previous treatment with Tarceva™, Iressa™, Rapamune™, temsirolimus or everolimus.
* Untreated metastasis to the central nervous system.
* Previous solid organ, bone marrow or stem-cell transplant.
* Known AIDS or HIV infection.
* Symptomatic or poorly controlled chronic heart failure.
* Chronic renal failure requiring dialysis on a regular basis.
* Chronic liver failure.
* Serum aspartate aminotransferase (AST), Alanine Aminotransferase (ALT), alkaline phosphatase or bilirubin >1.5 x the upper limit of normal for the local laboratory.
* Pregnant or breast-feeding women.
* Other invasive malignant diseases within 5 years (other than squamous or basal cell carcinoma of the skin).
* Inability to provide informed consent
* Any other serious and/or unstable medical, psychiatric, or other condition considered by the P.I. to preclude safe or reasonably compliant participation in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Flaig, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

REFERENCES:
- [Background] Gemmill RM, Zhou M, Costa L, Korch C, Bukowski RM, Drabkin HA. Synergistic growth inhibition by Iressa and Rapamycin is modulated by VHL mutations in renal cell carcinoma. Br J Cancer. 2005 Jun 20;92(12):2266-77. doi: 10.1038/sj.bjc.6602646. PMID 15956968

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase II, single-arm, single-institution trial. A total of 25 patients were enrolled between July 2006 and March 2008 from University of Colorado Cancer Center.
Pre-assignment Details: Patients with previous treatment with erlotinib, gefitinib, sirolimus, temsirolimus or everolimus, untreated central nervous system metastasis, renal failure requiring dialysis or significant liver dysfunction were excluded from the trial.
Groups:
- Erlotinib and Sirolimus: Erlotinib (Tarceva) therapy was started at 150 mg by mouth daily from day 1 to be taken at least 1 hour before or 2 hours after a meal. Sirolimus was initiated on day 8 (D8) with a loading dose of 6mg by mouth, followed by a daily dose of 2mg by mouth, on the basis of the product prescribing information for low-to-moderate immunologic risk renal transplant patients.
Period: Overall Study
Arm/Group | Erlotinib and Sirolimus
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: It was calculated that 25 participants will provide 80% power to detect an improvement in progression-free survival from 12 to 24 weeks in a pretreated population of renal cell carcinoma patients.
Arm/Group | Erlotinib and Sirolimus
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 60 [47 to 73]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Time to progression was defined as the time from beginning of therapy until disease progression or death. For subjects who had not progressed at the time of statistical analysis, progression-free survival was censored at the date of their last tumor assessment. Kaplan-Meier method was used to estimate median progression-free survival. Progression was defined as radiographic progression according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria (year 2000 version), non-compliance in obtaining scans, unequivocal clinical progression or the initiation of another medication for the treatment of renal cell carcinoma.
Time Frame: Physical exam assessments were performed every 4 weeks during the treatment phase. Survival follow-up information was collected every 4 months following the termination visit until death, loss to follow-up, or study termination up to 275 weeks.
Population: Per protocol analysis was used and 25 participants that were enrolled in the study were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Erlotinib and Sirolimus
Number analyzed (Participants) | 25
Weeks | 12 [5.9 to 18.1]

2. Secondary Outcome: Overall Survival
Description: For all subjects who had not died at the time of statistical analysis, duration of survival will was censored at the date of last contact. Kaplan-Meier methodology was used to estimate the magnitude of the treatment effect as described for progression-free survival.
Time Frame: Survival follow-up information was collected every 4 months following the termination visit until death, loss to follow-up, or study termination up to 275 weeks.
Population: Per protocol analysis was used and 25 participants that were enrolled in the study were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Erlotinib and Sirolimus
Number analyzed (Participants) | 25
Weeks | 40 [0 to 85.7]

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the period of active therapy up to 4 weeks.
Description: Monitoring included patient interview, physical exam, routine laboratory tests (even in absence of symptoms) and appropriate work-up of any new symptoms or laboratorial abnormalities.
Arm/Group | Erlotinib and Sirolimus
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib and Sirolimus (N=25)
Chest pain (Musculoskeletal and connective tissue disorders) | 1
Hospitalization (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib and Sirolimus (N=25)
Rash (Skin and subcutaneous tissue disorders) | 24
Dry skin (Skin and subcutaneous tissue disorders) | 8
Pruritis/pain (Skin and subcutaneous tissue disorders) | 6
Anaemia (Blood and lymphatic system disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 12
Anorexia (Gastrointestinal disorders) | 9
Mucositis (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 8
Hypoalbuminaemia (Blood and lymphatic system disorders) | 12
Elevated creatinine (Blood and lymphatic system disorders) | 10
Hypertriglyceridaemia (Blood and lymphatic system disorders) | 9
Hypophosphataemia (Blood and lymphatic system disorders) | 7
Fatigue (General disorders) | 11
Pain (General disorders) | 7
Chills/cold intolerance (General disorders) | 6
Weight loss (General disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 7
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Decreased left ventricular ejection fraction (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Anuria (Cardiac disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Haemorrhage/bleeding other (Respiratory, thoracic and mediastinal disorders) | 6

LIMITATIONS AND CAVEATS:
One limitation of this study was the lack of von Hippel-Lindau (VHL) mutational status assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes